CLINICAL TRIAL: NCT00019604
Title: The Use of Radiofrequency Ablation to Treat Hepatic Neoplasms
Brief Title: Radiofrequency Ablation in Treating Patients With Unresectable Primary or Metastatic Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator left the institution.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Caryn Steakley, R.N., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990025; 99-C-0025; CDR0000066875; NCT00001795 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Liver Cancer; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; liver metastases; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy; Radiofrequency Ablation; High-Energy Shock Waves; Fluorodeoxyglucose F18; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency ablation in liver cancer (Experimental): This trial is designed to gain experience with the use of ablation devices with liver tumors. Radiofrequency ablation is a procedure that heats tumors to several degrees above body temperature and may kill tumor cells.
  Interventions: Procedure: computed tomography; Procedure: magnetic resonance imaging; Procedure: positron emission tomography; Procedure: radiofrequency ablation; Procedure: radionuclide imaging; Procedure: ultrasound imaging; Radiation: fludeoxyglucose F 18 (FDG-PET); Radiation: gadopentetate dimeglumine

INTERVENTIONS:
Procedure: computed tomography — Scan to assess the effects of ablation.
Procedure: magnetic resonance imaging — Imaging used to assess the effects of this ablative therapy on tumor vascular density.
Procedure: positron emission tomography — Physiology based method of imaging disease based on uptake and metabolism of radiopharmaceutical by the tissues.
Procedure: radiofrequency ablation — Radiofrequency ablation uses saline infusion into and out of needle/electrode through a closed system. More energy may be deposited without tissue-charring or gas vaporization.
Procedure: radionuclide imaging — Imaging following injection of a radioactive material.
Procedure: ultrasound imaging — An ultrasound (e.g. sound waves) is used to identify the lesion and needle placement.
Radiation: fludeoxyglucose F 18 (FDG-PET) — FDG PET scans rely on metabolic changes to evaluate response to therapy.
Radiation: gadopentetate dimeglumine — Food and Drug Administration approved contrast agent.

SUMMARY:
RATIONALE: Radiofrequency ablation is a procedure that heats tumors to several degrees above body temperature and may kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiofrequency ablation in treating patients who have unresectable primary or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the nature and duration of response of patients with primary or metastatic liver neoplasms, who are not candidates for surgical resection, treated with radiofrequency interstitial tissue ablation.
* Evaluate the ability of dynamic magnetic resonance imaging (MRI) to assess the effects of this therapy on tumor blood flow and tumor vascular density in these patients.
* Determine the ability of positron emission tomography with fludeoxyglucose F 18 (FDG-PET) to monitor response after treatment with this therapy in these patients.
* Compare FDG-PET results with computed tomography (CT) scan, biopsy, and serum marker results in patients treated with this therapy.
* Compare the performance of FDG-PET with CT scan and MRI, in terms of their ability to assess the efficacy of this therapy in these patients.

OUTLINE: Lesions are targeted by ultrasound and then radiofrequency ablation needles are inserted into the lesions and heated to a target temperature greater than 60 degrees C for 15 minutes, though exposure time may vary depending on temperatures achieved. To achieve a 1 cm margin of ablated tissue around each lesion, multiple ablation courses may be performed, depending on the size of the lesions and the time required to complete the treatment.

Patients undergo magnetic resonance imaging with gadopentetate dimeglumine contrast, CT scan, ultrasound, and positron emission tomography with fludeoxyglucose F 18 at baseline, 6 weeks, every 3 months for 1 year, and then every 6 months for 2 years.

Patients are followed at 6 weeks, every 3 months for 1 year, and then every 6 months for 2 years or until evidence of recurrence.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or metastatic liver lesions

  * Not a candidate for surgical resection
* Must have six or fewer lesions and no single lesion greater than 7 cm in diameter
* Extrahepatic disease allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 50,000/mm^3
* Prothrombin time (PT) or partial thromboplastin time (PTT) no greater than 1.5 times control (except for therapeutically anticoagulated nonrelated medical conditions [e.g., atrial fibrillation])

Hepatic:

* Bilirubin no greater than 3.0 mg/dL

Renal:

* Creatinine no greater than 2.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No pacemakers, cerebral aneurysm clips, shrapnel injury, or implantable electronic devices
* No known uncontrollable serious reactions (e.g., anaphylaxis) to contrast agents used in this study
* Weight less than 136 kg

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Concurrent systemic therapy for extrahepatic disease is allowed only if begun prior to radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1998-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Libutti, MD, Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Ablation in Liver Cancer
Started | 44
Completed | 5
Not Completed | 39
Not completed — Death | 1
Not completed — Progressive disease | 23
Not completed — Refused treatment | 1
Not completed — Carcinoid tumor, not treatable | 1
Not completed — Going to have liver transplant | 1
Not completed — Move to a different study | 1
Not completed — Non compliant on systemic CH | 1
Not completed — Non compliant | 1
Not completed — Resectable disease | 1
Not completed — Started new chemo regimen | 1
Not completed — Pt going to immunotherapy study | 1
Not completed — Too much disease | 1
Not completed — Unable to evaluate | 1
Not completed — Details for other not available | 4

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.18 (13.19)
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Standard response criteria will be used to assess the CT (computed tomography) scan images on a lesion per lesion basis. Complete response is complete disappearance of the index lesion on followup scan when compared to the pretreatment images. Partial response is a decrease of 50% or greater in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images. Minor response is a decrease between 25% and 49% in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images. Stable disease is no change in the size of the treated lesion. Progressive disease is an increase of greater than 25% in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images.
Population: The time frame for this outcome measure is unknown; the investigator left the institution and there is no available data. We only have access available on 23 participants. We cannot comment on the others or verify because we do not have the data.
Measure: Number; unit: Participants
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 23
Participants
  Complete Response | 0
  Partial Response | 0
  Minor Response | 0
  Stable Disease | 0
  Progressive Disease | 23

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 9 years, 9 months
Population: NA is entered for the total number of participants with adverse events because it is unknown. Adverse event data is available but the format is uninterpretable.
Measure: Number; unit: Participants
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 44
Participants | NA — Adverse event data is available but the format is uninterpretable.

3. Secondary Outcome: Tumor Blood Flow
Description: Tumor blood flow was to be assessed by magnetic resonance imaging (MRI) and compared to data collected on baseline pretreatment images and other appropriate time points for changes in tumor microvascular density.
Time Frame: Baseline, 3 months, and 6 months following treatment
Population: This outcome measure was not analyzed because the investigator left the institution and the study never completed; all participants were taken off study.
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

4. Secondary Outcome: Tumor Vascular Density
Description: Tumor vascular density was to be assessed by magnetic resonance imaging (MRI) and compared to data collected on baseline pretreatment images and other appropriate time points for changes in tumor microvascular density. Patterns of MRI contrast uptake within tumors correlate with microvessel density.
Time Frame: Baseline, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With a Response Using Fludeoxyglucose (18F) - Positron Emission Tomography (FDG-PET) Following Radiofrequency Ablation (RFA)
Description: Response was to be evaluated by the standard response criteria. Complete response is the complete disappearance of the index lesion on follow-up scan when compared to the pretreatment images. Partial response is a decrease of 50% or greater in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images. Minor response is a decrease between 25% and 49% in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images. Stable disease is no change in the size of the treated lesion. Progressive disease is an increase of greater than 25% in the product of the perpendicular diameters of the measured lesion following treatment compared to the pretreatment images.
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

6. Secondary Outcome: Compare Fludeoxyglucose (18F) Positron-Emission Tomography (FDG-PET) Results With Computed Tomography (CT)
Description: Participants were to undergo FDG-PET scanning and CT scans to compare changes in size of metabolically active volume and standard uptake value (tumor metabolism).
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

7. Secondary Outcome: Compare Fludeoxyglucose (18F) Positron-Emission Tomography (FDG-PET) Results With Biopsies
Description: Participants were to undergo tissue biopsies of tumor to quantify changes in the tumor to see if the changes we see on the imaging studies are the same as the changes in the tumor.
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

8. Secondary Outcome: Compare Fludeoxyglucose (18F) Positron-Emission Tomography (FDG-PET) Results With Serum Markers
Description: Images obtained by the FDG-PET was to be processed for changes in measured parameters and quantified compared to serum markers at baseline and appropriate follow-up points.
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

9. Secondary Outcome: Compare the Performance of Fludeoxyglucose (18F) Positron-Emission Tomography to Computed Tomography and Magnetic Resonance Imaging With Respect to Their Ability to Assess the Effects of Radiofrequency Ablation on the Treatment of Hepatic Neoplasms
Description: Images obtained by the FDG-PET, MRI and CT was to be processed for changes in measured parameters and quantified compared to baseline (e.g., <median change, >median change in size on CT, computed by subtracting the baseline value from the value at the appropriate follow-up point).
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

10. Secondary Outcome: Evaluate the Ability of Fludeoxyglucose (18F) Positron-Emission Tomography (FDG-PET) to Monitor Response Following Radiofrequency Ablation (RFA)
Description: PET scan images was to be read by a physician experienced in the interpretation of whole body PET imaging. The region of interest was to be performed in any abnormal sites of uptake that is a candidate and or has been RFA ablated.
Time Frame: Baseline, 6 weeks, 3 months, and 6 months following treatment
Population: as for outcome 3
Arm/Group | Radiofrequency Ablation in Liver Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Number zero is entered for the total number of participants with adverse events because it is unknown. Adverse event data is available but it is uninterpretable, thus no Serious or Other adverse events are entered for this module.
Arm/Group | Radiofrequency Ablation in Liver Cancer
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Adverse event data is available but the format is uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No